CLINICAL TRIAL: NCT05131399
Title: Single Case Experimental Design (SCED) Comparing an Off-the-shelf Carbon Ankle Foot Orthosis (SPRYSTEP) Versus an off-the Shelf Standard Plastic Ankle Foot Orthosis in the Treatment of Walking Functional Impairment
Brief Title: Contribution of an Off-the-shelf Carbon Ankle Foot Orthosis (AFO) in the Management of Walking Functional Impairment
Acronym: DEFISTEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thuasne (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021-A02115-36
Record Dates: First submitted 2021-10-29; First posted 2021-11-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Neuropathy (Disorder)
Keywords: orthosis; functional walking impairment; foot drop; rehabilitation; GAS
MeSH Terms: conditions — Peroneal Neuropathies

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, interventional study, SCED design in ABAB introduction/withdrawal. The timing of the transition from one phase to the next will be randomized. The duration of each of the phases (A1, B1, A2, B2) will therefore be defined randomly, while maintaining a total duration of 12 weeks for each study schema.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-comparison (Experimental): Patients will be fitted with 2 types of ankle foot orthoses, alternately, divided into 4 phases, in the following order:
  Phase A1: Standard Plastic ankle foot orthosis Phase B1: carbon medical device ankle foot orthosis Phase A2: Standard Plastic ankle foot orthosis Phase B2: carbon medical device ankle foot orthosis Each patient is his own comparator. For all patients, the total duration of the study will be the same, and will correspond to 12 weeks.
  Interventions: Device: Phase A1; Device: Phase B1; Device: Phase A2; Device: Phase B2

INTERVENTIONS:
Device: Phase A1 — Plastic standard ankle foot orthosis
Device: Phase B1 — carbon medical device ankle foot orthosis
Device: Phase A2 — Plastic standard ankle foot orthosis
Device: Phase B2 — carbon medical device ankle foot orthosis

SUMMARY:
The objective of this study is to assess the superiority in achieving personal goals (set by the patient and the medical team) according to the GAS scale (Goal Attainment Scaling) while wearing the carbon medical device Ankle Foot Orthosis (AFO) compared to a standard plastic ankle foot orthosis.

DETAILED DESCRIPTION:
Foot drop is a symptom observed in various pathologies including neuro-muscular pathologies of peripheral or central origin. It is a walking disability, causing a deterioration in the patients autonomy and quality of life.

The current medical strategy focuses on various off-the-shelf or custom made devices, depending on the walking functional impairment and the characteristics of foot deformities.

The objective of this study is to assess the superiority in achieving personal goals (set by the patient and the medical team) according to the GAS scale (Goal Attainment Scaling) while wearing the carbon medical device ankle foot orthosis compared to a standard plastic ankle foot orthosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a foot levator muscles impairment (single or bilateral drop foot) and / or instability of the back of the foot, associated with a deficit of the triceps
* Patient with inability to stand on tip-toe on one foot
* Patient having signed a free and informed consent
* Patient affiliated or entitled to a social security scheme

Exclusion Criteria:

* Patient with fixed varus-equine foot
* Patient with an unstable skin condition (whether or not treated with additional treatment that may change the footwear)
* Patient with a a foot levator muscles impairment with a deficiency of the quadriceps and hamstrings (knee involvement)
* Patient with uncontrolled spasticity
* Patient for whom foot surgery is planned during the study
* Patient with one of the contraindications to the use of carbon medical device, indicated in the instructions for use
* Patient with one of the contraindications to the use of the standard plastic ankle foot orthosis, indicated in the instructions for use
* Patient with orthopedic comorbidities affecting the musculoskeletal system
* Pregnant woman
* Patient with major cognitive impairment incompatible with participation in a clinical trial
* Patient participating in another clinical investigation conducted to establish the compliance of a MD impacting the evaluation criteria
* Patient who cannot be followed for 12 weeks
* Vulnerable patient according to article L1121-6 of the public health code, persons subject to a measure of judicial protection or unable to consent freely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Comparison of the ability to achieve personal goals while wearing carbon or standard plastic ankle foot orthosis | 3 times a week during 12 weeks
  Personal goals achievement is evaluated via the Goal attainment scaling (GAS). Before starting the study, three personal objectives are defined according to patients needs and investigator review.
  Raw scores ranging from -3 (degradation) to +2 (maximum achievement of the objective) are defined:
  "-3" corresponding to degradation "-2" corresponding to the initial state "-1" corresponding to a partial objective achievement "0" corresponding to the total objective achievement "+1" corresponding to a better objective achievement "+2" corresponding to the maximum objective achievement. The GAS is filled 3 times a week during 12 weeks.

SECONDARY OUTCOMES:
Comparison of patients mobility while wearing carbon or standard plastic ankle foot orthosis | Visits V0 (Day 0), V1 (between week 2 and 3), V2 (between week 5 and 6), V3 (between week 8 and 9) and V4 (Week 12).
  Mobility is evaluated via staircase tests: Time (in minutes) to go up and down 10 steps
Comparison of patients walking perimeter while wearing carbon or standard plastic ankle foot orthosis | Visits V0 (Day 0), V1 (between week 2 and 3), V2 (between week 5 and 6), V3 (between week 8 and 9) and V4 (Week 12)
  Walking perimeter is evaluated via the Six-minute walk test (6MWT), that measures the distance (in meters) during a 6 minutes walk.
Comparison of patients fatigue while wearing carbon or standard plastic ankle foot orthosis | Visits V0 (Day 0), V1 (between week 2 and 3), V2 (between week 5 and 6), V3 (between week 8 and 9) and V4 (Week 12)
  Patient's fatigue perception is assessed by the patient via the Borg Rating of Perceived Exertion (RPE) scale following mobility and walking perimeter tests The effort rating is based on a scale of 6 to 20 (6, which is "no effort", to 20, which is "maximum effort").
Comparison of patients stability while wearing carbon or standard plastic ankle foot orthosis | Visits V0 (Day 0), V1 (between week 2 and 3), V2 (between week 5 and 6), V3 (between week 8 and 9) and V4 (Week 12)
  Patient's stability is assessed by 2 means:
  1. via the Timed Up and Go test : time (in seconds) to realize the test. The patient should stand up from a chair, walk a distance of three meters, turn around, then walk back to the chair and sit down. These tasks should be performed at a comfortable and safe speed.
  2. via the number of falls recorded during each phase and their context
Comparison of patients disability evolution according to the investigator while wearing carbon or standard plastic ankle foot orthosis | Visits V0 (Day 0), V1 (between week 2 and 3), V2 (between week 5 and 6), V3 (between week 8 and 9) and V4 (Week 12)
  Doctors' opinion on the Patients disability evolution is measured by the Clinical Global Impression - Improvement (CGI-I) questionnaire.
  The scale has 7 levels of answer from "very strongly improved" which is the better outcome (= 1 point) to "very strongly aggravated" which is the worst outcome (= 7 points) .Intermediate levels are: " Significantly improved "(= 2 points) ; " Slightly improved " (= 3 points) ; " No improvement " (=4 points) ; " Slightly worsen " (=5 points) ; " Seriously worsen" ( = 6 points).
  The highest score corresponds to the most impairment in quality of life.
Comparison of patients disability evolution according to the patient while wearing carbon or standard plastic ankle foot orthosis | Visits V0 (Day 0), V1 (between week 2 and 3), V2 (between week 5 and 6), V3 (between week 8 and 9) and V4 (Week 12)
  Patient's opinion on his disability evolution is measured by the Global Impression of Change (PCI-C).
  The scale has 7 levels from "no change or condition has got worsed"(worse outcome) to "a great deal better, and a considerable improvement that has made all the difference ( better outcome)". Intermediate levels are: "almost the same, hardly any change at all"; "a little better, but no noticeable change", "somewhat better, but the change has not made any real difference"; "moderately better, and a slight but noticeable change"; "better, and a definite improvement that has made a real and worthwhile difference.
Comparison of pain, gait and balance evolution according to the patient while wearing carbon or standard plastic ankle foot orthosis | Visits V0 (Day 0), V1 (between week 2 and 3), V2 (between week 5 and 6), V3 (between week 8 and 9) and V4 (Week 12)
  Pain level is measured by Visual Analogic Scale (VAS) completed by the patient : 0 corresponds to no pain (better outcome) and 10 to maximum pain (worst outcome).
  Natural gait and confidence in walking are measured by Visual Analogic Scale (VAS) completed by the patient : 0 corresponds to no natural gait or no confidence (worst outcome) and 10 to better natural gait and better confidence (better outcome).
  Balance is measured by Visual Analogic Scale (VAS) completed by the patient : 0 corresponds to no balance (worst outcome) and 10 to maximum balance (better outcome).
Comparison of tolerance of carbon and standard plastic ankle foot orthosis | Visits V0 (Day 0), V1 (between week 2 and 3), V2 (between week 5 and 6), V3 (between week 8 and 9) and V4 (Week 12)
  Tolerance is measured by reported adverse events. Number and type of serious and non-serious Adverse Device Effects (ADE) are reported.
Comparison of acceptability and compliance with carbon and standard plastic ankle foot orthosis | Visits V0 (Day 0), V1 (between week 2 and 3), V2 (between week 5 and 6), V3 (between week 8 and 9) and V4 (Week 12)
  Cumulative wearing time of the devices under study (indicated by a thermal button inserted into the device) is collected during each phase. Specific questions on compliance are also asked by the investigator to the patient during the various visits.
Patients satisfaction with carbon and standard plastic ankle foot orthosis | V4 at 12 weeks
  Patients satisfaction is evaluated at the end of phase B2 regarding the use of the study devices via the "Technology" part of the evaluation towards a technical aid questionnaire (8 questions) and a specific questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe THOUMIE, MD PhD, Principal Investigator — Hôpital Rothschild (Paris)
Locations (8):
- France (8):
  - Ch Les Capucins, Angers
  - Chu Dijon, Dijon
  - CH LAVAL, Laval
  - CHU Lille, Lille
  - centre Louis PIERQUIN, Nancy
  - CHU Nantes, Nantes
  - Hôpital Rothschild, Paris
  - CHU Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krasny-Pacini A, Evans J. Single-case experimental designs to assess intervention effectiveness in rehabilitation: A practical guide. Ann Phys Rehabil Med. 2018 May;61(3):164-179. doi: 10.1016/j.rehab.2017.12.002. Epub 2017 Dec 15. PMID 29253607
- [Background] Barreto LC, Oliveira FS, Nunes PS, de Franca Costa IM, Garcez CA, Goes GM, Neves EL, de Souza Siqueira Quintans J, de Souza Araujo AA. Epidemiologic Study of Charcot-Marie-Tooth Disease: A Systematic Review. Neuroepidemiology. 2016;46(3):157-65. doi: 10.1159/000443706. Epub 2016 Feb 6. PMID 26849231
- [Background] Gholizadeh H, Abu Osman NA, Eshraghi A, Ali S, Razak NA. Transtibial prosthesis suspension systems: systematic review of literature. Clin Biomech (Bristol). 2014 Jan;29(1):87-97. doi: 10.1016/j.clinbiomech.2013.10.013. Epub 2013 Oct 29. PMID 24315710
- [Background] Zucker DR, Ruthazer R, Schmid CH. Individual (N-of-1) trials can be combined to give population comparative treatment effect estimates: methodologic considerations. J Clin Epidemiol. 2010 Dec;63(12):1312-23. doi: 10.1016/j.jclinepi.2010.04.020. Epub 2010 Sep 22. PMID 20863658
- [Background] Spieler JF, Amarenco P. [Socio-economic aspects of stroke management]. Rev Neurol (Paris). 2004 Nov;160(11):1023-8. doi: 10.1016/s0035-3787(04)71139-x. French. PMID 15602344